CLINICAL TRIAL: NCT03993457
Title: Promoting Enhanced Pharmacotherapy Choice Through Immunomarkers Evaluation in Depression
Acronym: PRECISE-D
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: terminated during COVID due to inability to see participants in person.
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2019-0623
Record Dates: First submitted 2019-06-13; First posted 2019-06-20 (Actual); Results first posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Depression
Keywords: depression; mental health; mood disorders; major depressive episode; major depressive disorder; antidepressants; escitalopram; bupropion; depression treatment
MeSH Terms: conditions — Depression; Psychological Well-Being; Mood Disorders; Depressive Disorder, Major | interventions — Escitalopram; Bupropion

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two groups based on their CRP levels:
  * CRP less than 1
  * CRP greater than or equal to 1
  Participants within both groups will then be randomized to one of 2 groups, which is stratified by a CRP group:
  * CRP consistent antidepressant selection (medication will be prescribed based on CRP level)
  * CRP inconsistent antidepressant selection (medication will be prescribed in contradiction to CRP level)
Masking Description: Participant, care provider, investigator, and outcomes assessor will only be blinded to the participant's CRP levels and group assignment. However, the study is open label, meaning the participant, care provider, investigator, and outcomes assessor will know what medication the participant is taking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- CRP<1, CRP consistent antidepressant selection (Other): Participants with CRP<1 will be prescribed escitalopram
  Interventions: Drug: Escitalopram
- CRP> or equal to 1, CRP consistent antidepressant selection (Other): Participants with CRP> or equal to 1 will be prescribed bupropion XL
  Interventions: Drug: Bupropion
- CRP<1, CRP inconsistent antidepressant selection (Other): Participants with CRP< 1 will be prescribed bupropion XL
  Interventions: Drug: Bupropion
- CRP> or equal to 1, CRP inconsistent antidepressant selection (Other): Participants with CRP> or equal to 1 will be prescribed escitalopram
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram will be started at 5 mg/day during the first week of treatment. The dose will then be increased to 10mg/day, and can be increased to 20 mg/day. Dose can be decreased to 5 mg by clinician discretion such as to increase tolerability or better manage side-effects. 5 mg will be the lowest dose allowed in the study.
  Other Names: Lexapro
  Arms: CRP<1, CRP consistent antidepressant selection; CRP> or equal to 1, CRP inconsistent antidepressant selection
Drug: Bupropion — Bupropion-XL will be started at 150 mg/day and increased to 300 mg/day after one week. This dose can be increased to 450 mg/day (divided in 2 doses) at Week 2 or later. Clinicians may opt to titrate bupropion-XL in a slower fashion in cases that might increase tolerability or better manage side-effects. 150 mg will be the lowest dose allowed in the study.
  Other Names: Wellbutrin XL
  Arms: CRP<1, CRP inconsistent antidepressant selection; CRP> or equal to 1, CRP consistent antidepressant selection

SUMMARY:
PRECISE-D is a single site, randomized, open label 8-week clinical trial that will enroll 70 participants to evaluate if the level of inflammation in our body can predict how we will respond to antidepressants. C-reactive protein (CRP) is a substance in the body that is associated with inflammation. Previous research has suggested that people with high CRP (i.e., high inflammation levels) tend to have greater improvement of depressive symptoms with an antidepressant called bupropion, while individuals with low CRP (i.e., low inflammation levels) appear to have more benefit from selective serotonin reuptake inhibitors antidepressants (SSRI), such as escitalopram. However, it is not completely clear if CRP can predict your response to these two antidepressants.

Participants will undergo a screening visit that includes a physical exam, overall health evaluation, assessment of mental health history, and a toxicology and pregnancy test. Once screening is complete, participants will be randomized to one of two groups that will determine whether their CRP levels will be used to select which antidepressant they will receive. Participants will then complete 4 follow up visits at weeks 2, 4, 6, and 8. A follow-up phone call from the study team will occur at week 12.

DETAILED DESCRIPTION:
PRECISE-D is a single site, randomized, open label 8-week clinical trial that will enroll 70 participants. Participants will be asked to attend approximately 5 visits with the researchers or study staff.

The screening process will take approximately 2 hours, and will include a physical examination, toxicology and pregnancy test, as well as the completion of assessments. We will ask participants a series of questions regarding their general health, mental health history, and any medications they are currently taking. Additionally, some self-report questionnaires will be used as part of this process. The results of the screening exams, tests, and/or procedures will be reviewed to determine whether a participant will be allowed to continue in the study. In the event that there are questions about a participant's eligibility or screening procedures are remaining, the screening visit may be conducted over 2 visits.

Once eligibility is determined, the baseline visit (Week 0) will be completed. This visit will last approximately 1 hour and 15 minutes and will include the following:

* Bloodwork: We will obtain levels of CRP and other inflammatory substances. We will also examine electrolytes, kidney function, thyroid function, lipid panel, blood cell count, and other tests of general health.
* Self-Report Questionnaires: Participants will complete 8 questionnaires. These include questions about mental health and mood. The questionnaires range from 5 to 20+ items.
* Cognitive tests: We will examine the participant's attention, memory, and cognition using a series of computerized assessments.

Participants will be assigned to a study group based on their CRP level: CRP less than 1 (low CRP), or CRP greater than or equal to 1 (high CRP). Within this group assignment, participants will then be randomized, or assigned by chance (like flipping a coin), to one of 2 study groups:

• CRP consistent antidepressant selection (medication will be prescribed based on participant's CRP level).

If CRP less than 1, participant will be prescribed escitalopram. If CRP greater than or equal to 1, participant will be prescribed bupropion XL.

• CRP inconsistent antidepressant selection (medication will be prescribed in contradiction to participant's CRP level) If CRP less than 1, participant will be prescribed bupropion XL. If CRP greater than or equal to 1, participant will be prescribed escitalopram.

In each group participants will receive either escitalopram or bupropion XL.

* 1 tablet of 150 mg of bupropion-XL per day (initial dose). The dose will be increased to 300mg per day after the first week, and may be increased up to 450 mg/per day if deemed necessary by the clinician.
* 1 tablet of 5 mg of escitalopram per day (initial dose). The dose will be increased to 10 mg per day after the first week, followed by an additional increase to 20 mg/day if deemed necessary by clinician.

Participants and study doctors will know which medication is being used, but not which group the participant is in; that is, participants and study doctors will not know the participant's CRP levels nor whether the medication assignment is consistent with CRP levels. The dose of the medication may be adjusted up or down during the study to improve effects of the medication or reduce possible side effects. Dose changes will be made based on how the participant is feeling and any side effects.

Participants will then complete a clinical visit at Week 2, 4, and 6. These visits will last approximately 1 hour and 15 minutes, and will include the following:

* Clinical Evaluation: a psychiatrist will check the participant's vital signs and assess their overall wellbeing. Symptom changes, side effects, and adherence to treatment will be evaluated. Medication dosage adjustments will be made as necessary.
* Self-Report Questionnaires

The final clinical visit will occur at week 8. This visit will be the last in person visit and will last approximately 1 hour and 45 minutes. The following will be completed

* Clinical Evaluation
* Self-Report Questionnaires
* Cognitive tests
* Bloodwork
* Pregnancy test (if you are a female able to become pregnant)

After study completion, participants who wish to remain on treatment will be given a four week supply of study drug while they transition care.

Additionally, a remote follow up assessment will be done at Week 12. Participants will be contacted via phone to complete a series of questionnaires. Additionally, they will receive a series of self reports via email. Paper forms will be also available at the Center for Depression Research and Clinical Care if the participant prefers to answer them on paper or don't have access to an email.

The self-report questionnaires, study evaluations, and assessment of CRP levels and additional inflammatory substances in this study are designed for research, not for medical purposes. Even though the researchers are not specifically looking at blood to find a medical problem, participants will be notified if any abnormal results are identified.

Participants will also have the option to participate in a Finger Prick Blood CRP substudy that will compare CRP results based on the blood source: venous blood obtained via venipuncture and capillary blood obtained via finger prick. A few drops of capillary blood will be collected via finger prick once during the study at week 0 (screening/baseline). We will compare the finger prick results to the results obtained from venipuncture at the same visit.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ages 18-65
* Current diagnosis of Major Depressive Disorder
* Able to read, speak, and understand English

Exclusion Criteria:

* Antidepressant use within the last 8 weeks
* Active infection or uncontrolled autoimmune disease
* Currently on oral corticosteroids or active immune suppressive therapy (methotrexate, cyclosporine, anti-cytokines medications, etc).
* Current diagnosis of uncontrolled HIV, hepatitis C or significant immunodeficiency
* Alcohol or substance use disorder
* Positive urine drug test for illicit substances or substances used out of the context of prescription
* Cognitively unable to give informed consent
* Pregnant or breastfeeding women, women of childbearing potential who are not using an accepted means of birth control, or women with a positive urine pregnancy test
* History of seizure disorder
* Previous significant adverse reaction to escitalopram or bupropion
* History of non-response to adequate doses of escitalopram or bupropion XL
* Current use of concomitant psychotropic agents (anticonvulsants, benzodiazepines, hypnotics, opiates, triiodothyronine (T3), modafinil, psychostimulants, buspirone, melatonin, folate, l-methylfolate, s-adenosyl methionine, lithium) not on the same dose for at least four weeks prior to study entry or who do not agree to continue at the same dose during the acute phase of the study.
* Lifetime history of bipolar disorder, schizophrenia, schizoaffective disorder or other psychotic disorder
* Current anorexia nervosa or bulimia nervosa
* Suicidal ideation of the degree that, in the opinion of the evaluating clinician, participation in the study would place them at significantly increased risk of suicide
* Unstable medical issues of such degree that, in the opinion of the evaluating clinician, participation in the study would place them at significant risk of a serious adverse event

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar H Trivedi, MD, Principal Investigator — UTSW
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CRP<1, CRP Consistent Antidepressant Selection | CRP> or Equal to 1, CRP Consistent Antidepressant Selection | CRP<1, CRP Inconsistent Antidepressant Selection | CRP> or Equal to 1, CRP Inconsistent Antidepressant Selection
Started | 4 | 2 | 1 | 4
Completed | 4 | 2 | 1 | 2
Not Completed | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- CRP> or Equal to 1, CRP Consistent Antidepressant: Participants with CRP> or equal to 1 will be prescribed bupropion XL
  Bupropion: Bupropion-XL will be started at 150 mg/day and increased to 300 mg/day after one week. This dose can be increased to 450 mg/day (divided in 2 doses) at Week 2 or later. Clinicians may opt to titrate bupropion-XL in a slower fashion in cases that might increase tolerability or better manage side-effects. 150 mg will be the lowest dose allowed in the study.
- Total: Total of all reporting groups
Arm/Group | CRP<1, CRP Consistent Antidepressant Selection | CRP> or Equal to 1, CRP Consistent Antidepressant | CRP<1, CRP Inconsistent Antidepressant Selection | CRP> or Equal to 1, CRP Inconsistent Antidepressant Selection | Total
Number analyzed (Participants) | 4 | 2 | 1 | 4 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 1 | 4 | 11
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.3 (15.2) | 33.5 (9.2) | 25 (0) | 25.7 (10.8) | 33.8 (13.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 2 | 1 | 1 | 2 | 6
  Gender: Male | 2 | 1 | 0 | 1 | 4
  Gender: Unknown/Not Reported | 0 | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 2 | 6
  Not Hispanic or Latino | 3 | 0 | 0 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1
  White | 2 | 1 | 0 | 3 | 6
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 1 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of CRP-consistent Antidepressant Selection Versus CRP-inconsistent Antidepressant Selection on Remission Rates in Patients With MDD.
Description: The primary study endpoint will be remission rates based on the 16-items Quick Inventory of Depressive Symptomatology, Self-Report (QIDS-SR), which will be extracted from the 30-item Inventory of Depressive Symptomatology (IDS-SR). The QIDS-SR score ranges from 0-27. A score of 5 or less represents remission.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | CRP<1, CRP Consistent Antidepressant Selection | CRP> or Equal to 1, CRP Consistent Antidepressant Selection | CRP<1, CRP Inconsistent Antidepressant Selection | CRP> or Equal to 1, CRP Inconsistent Antidepressant Selection
Number analyzed (Participants) | 4 | 2 | 1 | 4
Participants | 3 | 1 | 1 | 2

2. Primary Outcome: Efficacy of CRP-consistent Antidepressant Selection Versus CRP-inconsistent Antidepressant Selection on Improving Social and Occupational Functioning.
Description: Improvement in social and occupational functioning will be measured with the 5-item self-administered Work and Social Adjustment Scale (WSAS). The WSAS total score ranges from 0-40. Lower scores are better.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CRP<1, CRP Consistent Antidepressant Selection | CRP> or Equal to 1, CRP Consistent Antidepressant Selection | CRP<1, CRP Inconsistent Antidepressant Selection | CRP> or Equal to 1, CRP Inconsistent Antidepressant Selection
Number analyzed (Participants) | 4 | 2 | 1 | 2
score on a scale | -17.3 (8.0) | -24.4 (20.3) | -18.0 (0) | -23.5 (0.7)

3. Primary Outcome: Adverse Antidepressant Treatment Effects on CRP-consistent Antidepressant Selection Versus CRP-inconsistent Antidepressant Selection
Description: Side effects will be assessed using the 3-item self-administered Frequency, Intensity, and Burden of Side Effects (FIBSER). Each item is scored on a scale from 0-6. Items 1 and 2 (Frequency & Intensity respectively) are to provide information to the clinician, but they are not used in the scoring.The score that is used comes only from Item 3 - Burden. Lower scores represents lower burden.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CRP<1, CRP Consistent Antidepressant Selection | CRP> or Equal to 1, CRP Consistent Antidepressant Selection | CRP<1, CRP Inconsistent Antidepressant Selection | CRP> or Equal to 1, CRP Inconsistent Antidepressant Selection
Number analyzed (Participants) | 4 | 2 | 1 | 2
score on a scale | .25 (.5) | 0 (0) | 0 (0) | 0 (0)

4. Secondary Outcome: Optional Sub-study. Validity and Reliability of Capillary Blood CRP Measurement
Description: Capillary blood CRP levels will be compared with those obtained using venous blood obtained via venipuncture. Outcome will be number of participants whose capillary blood CRP levels and venous blood CRPT levels match in terms of <1 vs. >=1.
Time Frame: Baseline
Population: Some participants did not have a venous blood CRP conducted.
Measure: Count of Participants; unit: Participants
Arm/Group | CRP<1, CRP Consistent Antidepressant Selection | CRP> or Equal to 1, CRP Consistent Antidepressant Selection | CRP<1, CRP Inconsistent Antidepressant Selection | CRP> or Equal to 1, CRP Inconsistent Antidepressant Selection
Number analyzed (Participants) | 2 | 0 | 1 | 4
Participants | 2 | 0 | 1 | 4

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | CRP<1, CRP Consistent Antidepressant Selection | CRP> or Equal to 1, CRP Consistent Antidepressant Selection | CRP<1, CRP Inconsistent Antidepressant Selection | CRP> or Equal to 1, CRP Inconsistent Antidepressant Selection
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 1/2 | 1/1 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRP<1, CRP Consistent Antidepressant Selection (N=4) | CRP> or Equal to 1, CRP Consistent Antidepressant Selection (N=2) | CRP<1, CRP Inconsistent Antidepressant Selection (N=1) | CRP> or Equal to 1, CRP Inconsistent Antidepressant Selection (N=4)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — fall leading to lower back pain
worsening anxiety symptoms (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — including restlessness, vivid dreams
night insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — since starting 300mg dose
headaches (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
mouth sores (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
epigastric pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
heart palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
heartburn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
upset stomach (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT03993457/Prot_000.pdf